CLINICAL TRIAL: NCT00405535
Title: Adjunctive Glycine for Obsessive Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Collaborators: Obsessive Compulsive Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04I/C06
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Obsessive Compulsive Disorder
Keywords: OCD; Obsessive Compulsive Disorder; Glycine
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Glycine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): glycine powder
  Interventions: Drug: glycine
- B (Placebo Comparator): placebo powder
  Interventions: Other: placebo

INTERVENTIONS:
Drug: glycine
  Arms: A
Other: placebo
  Arms: B

SUMMARY:
The purpose of this study is to determine whether individuals with obsessive compulsive disorder who will take a preparation of the amino acid glycine in addition to their current treatment, may experience improvement in their symptoms.

DETAILED DESCRIPTION:
Individuals with obsessive compulsive disorder (OCD) often find inadequate relief, even with the best of currently available treatments. Some evidence suggests the the neurotransmitter glutamate may be a useful target for new treatments for OCD. The amino acid glycine, if given orally in adequate dosages, can have specific effects on one particular glutamate receptor molecule in the brain, that might be helpful with OC symptoms. This randomized, double-blind protocol will have study participants who suffer with OCD take either a glycine preparation or placebo for 12 weeks. Clinical measures (e.g., Y-BOCS, NIMH-OC) will be recorded at each visit to determine whether those taking the glycine experience clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OCD present for at least 1 year
* Male or female, age 18 to 65
* Stable medication regimen for 12 weeks prior to study entry
* at least moderately severe OC symptoms

Exclusion Criteria:

* Active substance use disorder within the last 6 months
* Comorbid schizophrenia, schizoaffective disorder, bipolar disorder, tic disorder, Tourette Disorder, schizotypal personality disorder
* Hoarding as the principal OCD symptom
* Insulin-dependent diabetes mellitus
* Pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-06; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Y-BOCS (Yale-Brown Obsessive Compulsive Scale) | 12 weeks after baseline

SECONDARY OUTCOMES:
NIMC-OC scale | 12 weeks after baseline
CGI-Improvement | 12 weeks after baseline
QLS(Quality of Life Scale) | 12 weeks after baseline
Sheehan Disability Scale | 12 weeks after baseline

CONTACTS AND LOCATIONS:
Overall Officials: William M Greenberg, MD, Principal Investigator — Nathan Kline Institute for Psychiatric Research
Locations (1):
- The Nathan Kline Institute for Psychiatric Research, Orangeburg, New York, United States

REFERENCES:
- [Derived] Greenberg WM, Benedict MM, Doerfer J, Perrin M, Panek L, Cleveland WL, Javitt DC. Adjunctive glycine in the treatment of obsessive-compulsive disorder in adults. J Psychiatr Res. 2009 Mar;43(6):664-70. doi: 10.1016/j.jpsychires.2008.10.007. Epub 2008 Nov 30. PMID 19046587